CLINICAL TRIAL: NCT06076902
Title: Patch Study: a Single-center, Prospective, Single-blind, Randomized, Two-arm Controlled Study of Outcomes Following Synthetic Polyester Patch-augmented Rotator Cuff Repair
Brief Title: Patch Study (Patch-augmented Rotator Cuff Repair)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Spital Thurgau AG (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ProjectID 2023-00238
Record Dates: First submitted 2023-09-18; First posted 2023-10-11 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Rotator Cuff Tears
Keywords: Rotator Cuff Repair
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single blind study in which only patients will not be aware of treatment (with or without rotator cuff augmentation with polyester patch)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment group with patch augmentation (Experimental): Arthroscopic rotator cuff reconstruction using fixation with anchors augmented with a synthetic polyester patch
  Interventions: Device: Arthroscopic rotator cuff reconstruction using fixation with anchors augmented with a synthetic polyester patch (Pitch-Patch Tissue Reinforcement Device))
- Comparison group without patch augmentation (Active Comparator): Arthroscopic rotator cuff reconstruction using fixation with anchors and no augmentation with a synthetic polyester patch
  Interventions: Device: Arthroscopic rotator cuff reconstruction using fixation with anchors augmented without a synthetic polyester patch

INTERVENTIONS:
Device: Arthroscopic rotator cuff reconstruction using fixation with anchors augmented with a synthetic polyester patch (Pitch-Patch Tissue Reinforcement Device)) — The Pitch-Patch is a single-use device intended to reinforce the rotator cuff following or during repair by sutures or suture anchors where weakness exists in the soft tissue.
  Other Names: Pitch-Patch Tissue Reinforcement Device (version model number 102-1090)
  Arms: Treatment group with patch augmentation
Device: Arthroscopic rotator cuff reconstruction using fixation with anchors augmented without a synthetic polyester patch — Arthroscopic rotator cuff reconstruction using fixation with anchors and no augmentation with a synthetic polyester patch.
  Arms: Comparison group without patch augmentation

SUMMARY:
This single-center, prospective, randomized controlled study will compare patients allocated to two treatment arms who are undergoing surgery to repair rotator cuff tears: (1) arthroscopic rotator cuff reconstruction using fixation with anchors augmented with a synthetic polyester patch, and (2) arthroscopic rotator cuff reconstruction using fixation with anchors and no augmentation with a synthetic polyester patch. The primary objective is to compare complications (primarily retear rates) and the secondary objective is to compare mid- and long-term clinical and radiological outcomes using standard orthopedic assessments, such as the subjective shoulder value and the Constant-Murley score.

DETAILED DESCRIPTION:
This single-center, prospective, randomized controlled study will compare patients allocated to two treatment arms who are undergoing surgery to repair rotator cuff tears: (1) arthroscopic rotator cuff reconstruction using fixation with anchors augmented with a synthetic polyester patch, and (2) arthroscopic rotator cuff reconstruction using fixation with anchors and no augmentation with a synthetic polyester patch. The primary objective is to compare complications (primarily retear rates) and the secondary objective is to compare mid- and long-term clinical and radiological outcomes using standard orthopedic assessments, such as the subjective shoulder value and the Constant-Murley score.

The Pitch-Patch is a single-use synthetic polyester patch (Pitch-Patch, neoligamentsTM, Leeds, UK) intended to reinforce the rotator cuff following or during repair by sutures or suture anchors where weakness exists in the soft tissue. The surgical group will be randomly assigned, and each group will include 150 patients. After surgery, patients will be followed for two years and undergo clinical and radiological assessments.

The main research question to be answered by this investigation is whether synthetic patch augmentation can significantly improve outcomes in patients with rotator cuff tears from either degenerative or traumatic origins versus patients with no patch augmentation.

ELIGIBILITY:
Inclusion Criteria:

* Adults with massive rotator cuff tear
* Tear must affect at least two tendons
* Primary surgery only
* Origin of tear can be either degenerative or traumatic
* German language speaking

Exclusion Criteria:

* Fatty infiltration grade 4 (according to Goutallier)
* Bilateral tears
* Cases of arthritis or severe osteoarthritis
* Structural or pathological condition of the bone or soft tissue that could impair healing
* Unable or unwilling to restrict activities to prescribed levels or follow rehabilitation guidelines
* Unable or unwilling to give consent (language barrier or cognitive impairment)
* Unwilling or unable to be assessed at 1- and 2-year follow-up assessment visits

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-04-06 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Rotator cuff retear rate | Up to two years postoperative
  Occurence of retear following rotator cuff reconstruction to treat massive tear (measured using radiological imaging/ultrasound)

SECONDARY OUTCOMES:
Complication rate (adverse event greater than grade 2) | Up to two years postoperative
  Development of postoperative complications following rotator cuff reconstruction to treat massive tear
Pain levels | Preoperative and postoperative (6 weeks, 3 months, 1- and 2-year follow-up visits)
  During clinical assessments, patient reported pain levels will be measured using visual analogue scale (VAS); scale 0 (low) to 15 (high)
Healing rate | 6-week and 1-year exams (postoperative)
  Using radiological imaging (ultrasound), healing of the rotator cuff tear will be monitored over time
Range of motion | Preoperative and postoperative (6 weeks, 3 months, 1- and 2-year follow-up visits)
  Clinical assessments of healing using the range of motion will be compared over time

CONTACTS AND LOCATIONS:
Overall Officials: Florian Hess, MD, Principal Investigator — Spital Thurgau AG
Locations (1):
- Spital Thurgau AG, Frauenfeld, Thurgau, Switzerland